CLINICAL TRIAL: NCT05630352
Title: A MASTER PROTOCOL TO INVESTIGATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF BIVALENT BNT162b2 RNA-BASED VACCINE CANDIDATE(S) IN HEALTHY INFANTS AND CHILDREN
Brief Title: A Study to Learn About Bivalent COVID-19 RNA Vaccine Candidate(s) in Healthy Infants and Children
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Bivalent vaccine no longer epidemiologically relevant.
Sponsor: BioNTech SE (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: C4591023
Record Dates: First submitted 2022-11-22; First posted 2022-11-29 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: COVID-19
Keywords: SARS-CoV-2 infection; COVID-19; SARS-CoV-2 Virus; Severe Acute Respiratory Syndrome Coronavirus 2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Phase 1 open label sequential dose escalation study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dose level 1 (Experimental): Injection in the muscle at 0-, 8-, and 16-weeks.
  Interventions: Biological: Bivalent BNT162b2 (original/Omicron BA.4/BA.5) 3 microgram dose
- Dose level 2 (Experimental): Injection in the muscle at 0-, 8-, and 16-weeks
  Interventions: Biological: Bivalent BNT162b2 (original/Omicron BA.4/BA.5) 6 microgram dose
- Dose level 3 (Experimental): Infection in the muscle at 0-, 8- and 16- weeks
  Interventions: Biological: Bivalent BNT162b2 (original/Omicron BA.4/BA.5) 10 microgram dose
- Dose level 4 (Experimental): Injection in the muscle at 0-, 8- and 16- weeks
  Interventions: Biological: Bivalent BNT162b2 (original/Omicron BA.4/BA.5) 1 microgram dose

INTERVENTIONS:
Biological: Bivalent BNT162b2 (original/Omicron BA.4/BA.5) 3 microgram dose — Injection in the muscle
  Arms: Dose level 1
Biological: Bivalent BNT162b2 (original/Omicron BA.4/BA.5) 6 microgram dose — Injection in the muscle
  Arms: Dose level 2
Biological: Bivalent BNT162b2 (original/Omicron BA.4/BA.5) 10 microgram dose — Injection in the muscle
  Arms: Dose level 3
Biological: Bivalent BNT162b2 (original/Omicron BA.4/BA.5) 1 microgram dose — Injection in the muscle
  Arms: Dose level 4

SUMMARY:
The purpose of this clinical trial is to learn about the safety and immune responses of the study vaccine (called a bivalent BNT162b2 Omicron containing vaccine) in healthy infants and children. Sub study A of this clinical trial will test up to four different dose levels of the vaccine in infants who are under 6 months of age and have not previously received a coronavirus vaccination.

This will be a 3- dose primary series of the study vaccine with each dose separated by 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female participants 72 through 102 days of age, at the time of randomization (the day of birth is considered Day 1 of life).
2. Male or female participants born at greater than 32 weeks of gestation.

Exclusion Criteria:

1. Receipt of any nonstudy vaccine within 14 days, before study intervention administration (Dose 1 only).
2. Receipt of medications intended to prevent COVID-19.
3. Previous or current diagnosis of MIS-C (Multisystem Inflammatory Syndrome In Children).
4. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (e.g., anaphylaxis) to any component of the study intervention(s).
5. Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
6. Individuals with a history of autoimmune disease or an active autoimmune disease requiring therapeutic intervention.
7. Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
8. Other medical (e.g,. major known congenital malformation or serious chronic disorder such as seizures) or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study. Note: This includes both conditions that may increase the risk associated with study intervention administration or conditions that may interfere with the interpretation of study results.
9. Previous vaccination with any non-study coronavirus vaccine.
10. Individuals who receive treatment with immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids.
11. Receipt of blood/plasma products, immunoglobulin, or monoclonal antibodies (except palivizumab and hepatitis B immunoglobulin), from 60 days before study intervention administration, or receipt of any passive antibody therapy specific to COVID-19 from 90 days before study intervention administration, or planned receipt throughout the study.
12. Receipt of other study intervention within 28 days prior to study entry through and including 28 days after the last dose of study intervention, with the exception of non-Pfizer interventional studies for prevention of COVID-19, which are prohibited throughout study participation.
13. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members. Children or grandchildren who are direct descendants of investigator site staff or sponsor and sponsor delegate employees directly involved in the conduct of the study.

Ages: 72 Days to 102 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2025-01-06 (Estimated); Primary Completion 2026-07-13 (Estimated); Study Completion 2026-07-13 (Estimated)

PRIMARY OUTCOMES:
Substudy A - Percentage of participants reporting local reactions in each dose level | For 7 days following Dose 1, Dose 2, Dose 3
  Tenderness at the injection site, redness, and swelling as self-reported on electronic diaries.
Substudy A - Percentage of participants reporting systemic events in each dose level | For 7 days following Dose 1, Dose 2 and Dose 3
  Fever, decreased appetite, drowsiness, and irritability as self-reported on electronic diaries.
Substudy A - Percentage of participants reporting adverse events in each dose level | Dose 1 through 1 month after Dose 3
  As elicited by investigational site staff
Substudy A - Percentage of participants reporting serious adverse events in each dose level | Dose 1 through 6 months after Dose 3
  As elicited by investigational site staff

SECONDARY OUTCOMES:
Substudy A - Geometric mean titers elicited by prophylactic bivalent BNT162b2 at each dose level in COVID-19 vaccine-naïve participants < 6 months of age | At baseline (before Dose 1), 1 month after Dose 2, and 1 month after Dose 3
  As measured at the central laboratory
Substudy A - Geometric mean fold rise elicited by prophylactic bivalent BNT162b2 at each dose level in COVID-19 vaccine-naïve participants < 6 months of age | At baseline (before Dose 1), 1 month after Dose 2, and 1 month after Dose 3
  As measured at the central laboratory
Substudy A - Percentage of participants with seroresponse elicited by prophylactic bivalent BNT162b2 at each dose level in COVID-19 vaccine-naïve participants < 6 months of age | At baseline (before Dose 1), 1 month after Dose 2, and 1 month after Dose 3
  As measured at the central laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591023